CLINICAL TRIAL: NCT02809586
Title: Social Media Interventions to Reduce Alcohol Use Among Youth
Brief Title: Social Media Alcohol Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Maureen A Walton, Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: AA024175; R01AA024175 (NIH)
Record Dates: First submitted 2016-06-08; First posted 2016-06-22 (Estimated); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Drinking Behavior; Risky Drinking
Keywords: Alcohol; Teens; Young Adults; Social Media
MeSH Terms: conditions — Drinking Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- SMI + Incentives (Active Comparator): A Social Media + Incentives (SMI + I) condition
  Interventions: Behavioral: SMI + I
- SMI (Active Comparator): A Social Media Intervention (SMI) condition
  Interventions: Behavioral: SMI
- Control (No Intervention): An Attention-Control E-News (CONTROL) condition

INTERVENTIONS:
Behavioral: SMI + I — This 8-week social media based intervention consists of e-coaches delivering positive content to facilitate peer interaction. Participants will earn incentives for interaction during the intervention (8 weeks).
  Other Names: Social Media Intervention + Incentives
  Arms: SMI + Incentives
Behavioral: SMI — This 8-week social media based intervention consists of e-coaches delivering positive content to facilitate peer interaction. This group will NOT receive incentives for their participation in the secret group.
  Other Names: Social Media Intervention
  Arms: SMI

SUMMARY:
Social media provides frequent interaction with online social networks, increasing exposure to peer influences, which could affect alcohol use in negative or positive ways. The proposed study will recruit adolescents and emerging adults using social media ads, and conduct online screening, enrolling 975 risky drinkers in a randomized controlled trial comparing three conditions: 8-week Social Media Intervention + Incentives, 8-week Social Media Intervention Only, and an e-news attention control condition. These innovative design features will provide the critical next step in harnessing social media to reduce alcohol misuse, which could have enormous public health impact by altering the alcohol use trajectories of youth.

DETAILED DESCRIPTION:
The proposed study will recruit adolescents and emerging adults (ages 16-24) using social media ads and conduct online screening, enrolling 975 risky drinkers (i.e., using AUDIT-C screener) in a randomized controlled trial (RCT) comparing three conditions: 1) Social Media Intervention + Incentives (n=325), 2) Social Media Intervention Only (n=325), and 3) Attention Control E-News condition (n=325), with post baseline follow-up assessments at 3, 6, and 12 months. Interventions will include access for 8 weeks to unique, secret group pages facilitated by e-coaches (supervised by therapists), with dynamic content emphasizing reducing alcohol use/misuse as well as concomitant risk behaviors (other drug use based on co-ingestion and common motives for use).

ELIGIBILITY:
Inclusion Criteria:

Individuals will be eligible to participate if they are between the ages of 16 and 24 years and they have a Facebook account. Additionally, individuals will be eligible if they:

* Have a Past 3-month AUDIT-C score (see below) indicating that they meet criteria for at-risk drinking/alcohol misuse.

  * ages 16-17: ≥3 females and ≥4 males
  * ages 18-24: ≥4 females and ≥5 males

Exclusion Criteria:

* do not live in an area that the study is currently seeking participants from (i.e.- zip code not in area of active recruitment).
* under 16 years of age or over 24 years of age
* not Facebook account holder
* inability to give informed, voluntary consent

Ages: 16 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 955 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2020-06-25 (Actual); Study Completion 2020-06-25 (Actual)

PRIMARY OUTCOMES:
Change in Alcohol Consumption | 3-, 6-, and 12- months post baseline
  30-day Timeline Follow-Back (TLFB) will be used to assess alcohol consumption, binge drinking, quantity, and frequency of use.
Change in Alcohol Related Consequences | 3-, 6-, and 12- months post baseline
  Alcohol related consequences will be measured using the Young Adult Alcohol Consequences Questionnaire (YAACQ).

CONTACTS AND LOCATIONS:
Overall Officials: Maureen A Walton, MPH, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Florimbio AR, Coughlin LN, Bauermeister JA, Young SD, Zimmerman MA, Walton MA, Bonar EE. Risky Drinking in Adolescents and Emerging Adults: Differences between Individuals Using Alcohol Only versus Polysubstances. Subst Use Misuse. 2023;58(2):211-220. doi: 10.1080/10826084.2022.2152192. Epub 2022 Dec 20. PMID 36537360
- [Derived] Bonar EE, Bauermeister JA, Blow FC, Bohnert ASB, Bourque C, Coughlin LN, Davis AK, Florimbio AR, Goldstick JE, Wisnieski DM, Young SD, Walton MA. A randomized controlled trial of social media interventions for risky drinking among adolescents and emerging adults. Drug Alcohol Depend. 2022 Aug 1;237:109532. doi: 10.1016/j.drugalcdep.2022.109532. Epub 2022 Jun 11. PMID 35759874
- [Derived] Bonar EE, Souweidane MA, Blow FC, Bohnert ASB, Bauermeister JA, Young SD, Walton MA. High-intensity drinking among adolescent and emerging adult risky drinkers. Subst Abus. 2022;43(1):713-721. doi: 10.1080/08897077.2021.2007513. PMID 35100097
- [Derived] Bonar EE, Schneeberger DM, Bourque C, Bauermeister JA, Young SD, Blow FC, Cunningham RM, Bohnert AS, Zimmerman MA, Walton MA. Social Media Interventions for Risky Drinking Among Adolescents and Emerging Adults: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2020 May 13;9(5):e16688. doi: 10.2196/16688. PMID 32401225

DOCUMENTS (1):
  • Informed Consent Form (2019-12-11): https://cdn.clinicaltrials.gov/large-docs/86/NCT02809586/ICF_000.pdf